CLINICAL TRIAL: NCT01254409
Title: A Randomized, Double-Masked, Sponsor-Unmasked, Ascending Multiple Dose Study of the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of PRM-151 Administered Intravenously to Patients With Idiopathic Pulmonary Fibrosis
Brief Title: A Phase 1b Study of IV PRM151 in Patients With Idiopathic Pulmonary Fibrosis (IPF)
Acronym: PRM151F-12GL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WA42403; PRM151F-12GL (Other: Promedior, Inc.)
Record Dates: First submitted 2010-12-03; First posted 2010-12-06 (Estimated); Results first posted 2014-11-03 (Estimated); Last update posted 2022-04-20 (Actual); Status verified 2022-03

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: pulmonary, fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Pulmonary Fibrosis | interventions — PRM-151

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PRM-151 (Experimental): PRM-151 administered at escalating doses of 1, 5, and 10 mg/kg by 30 minute intravenous (IV) infusion days 1, 3, 5, 8 and 15.
  Interventions: Biological: PRM-151
- Placebo (Placebo Comparator): 0.9% saline administered by 30 minute IV infusion Days 1, 3, 5, 8, and 15.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: PRM-151 — Intravenous PRM-151 administered over 30 minutes on study days 1, 3, 5, 8, and 15 at doses of 1.0, 5.0, or 10.0 mg/kg.
  Arms: PRM-151
Other: Placebo — Intravenous 0.9% normal saline administered over 30 minutes on study days 1, 3, 5, 8, and 15.
  Arms: Placebo

SUMMARY:
The aims of the study are to assess safety, tolerability, the pharmacokinetic profile, and the pharmacodynamic profile of multiple doses of PRM-151 administered IV to IPF patients.

DETAILED DESCRIPTION:
Idiopathic pulmonary fibrosis (IPF) is a diffuse lung disease with a histological picture of usual interstitial pneumonia and a deteriorating clinical course. The prognosis is poor. Chronic alveolar inflammation with associated parenchymal remodeling is theorized to promote an ongoing abnormal fibrogenic repair response. Corticosteroids and immunomodulatory agents have not been shown to benefit IPF patients. Recently several published clinical studies have indicated a strong correlation between IPF severity and/or disease progression and the levels of specific plasma biomarker proteins related to epithelial cell health and extracellular matrix turnover.

PRM-151 is being developed for potential therapeutic uses to prevent, treat, and reduce fibrosis.

This study is the first intravenous multiple-dose study in humans, and will be conducted in patients with IPF. Patients will be randomized to receive either PRM-151 or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Men or women of non-childbearing potential aged 40 to 80 years at screening.
* Diagnosis of idiopathic pulmonary fibrosis (IPF) as determined by high resolution computerized tomography (HRCT) and pulmonary function tests.

Exclusion Criteria:

* History or presence of connective tissue disorder, tuberculosis (TB), cystic fibrosis, sarcoidosis, amyloidosis or other pulmonary disease except idiopathic pulmonary fibrosis (IPF).
* History or presence of chronic pulmonary obstructive disease, severe pulmonary hypertension, drug-induced pulmonary toxicity, other forms of idiopathic pneumonia, or interstitial lung diseases associated with environmental exposure medication or systemic disease.
* High resolution computerized tomography (HRCT) findings inconsistent with idiopathic pulmonary fibrosis(IPF).

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2011-03-29 (Actual); Primary Completion 2012-07-02 (Actual); Study Completion 2012-07-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Getsy, DMD, DO, Study Director — Hoffmann-La Roche
Locations (3):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Duke Clinical Research Unit, Durham, North Carolina
- Center for Human Drug Research, Leiden, Netherlands

REFERENCES:
- [Derived] van den Blink B, Dillingh MR, Ginns LC, Morrison LD, Moerland M, Wijsenbeek M, Trehu EG, Bartholmai BJ, Burggraaf J. Recombinant human pentraxin-2 therapy in patients with idiopathic pulmonary fibrosis: safety, pharmacokinetics and exploratory efficacy. Eur Respir J. 2016 Mar;47(3):889-97. doi: 10.1183/13993003.00850-2015. Epub 2016 Feb 11. PMID 26869678

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: 0.9% saline administered as a 30 minute IV infusion Days 1, 3, 5, 8 and 15
- PRM-151 1 mg/kg: PRM-151 1 mg/kg administered as a 30 minute IV infusion Days 1, 3, 5, 8 and 15
- PRM-151 5 mg/kg: PRM-151 5 mg/kg administered as a 30 minute IV infusion Days 1, 3, 5, 8 and 15
- PRM-151 10 mg/kg: PRM-151 10 mg/kg administered as a 30 minute IV infusion Days 1, 3, 5, 8 and 15
Period: Overall Study
Arm/Group | Placebo | PRM-151 1 mg/kg | PRM-151 5 mg/kg | PRM-151 10 mg/kg
Started | 6 | 6 | 5 | 4
Completed | 6 | 5 | 5 | 4
Not Completed | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All subjects enrolled in study
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | PRM-151 1 mg/kg | PRM-151 5 mg/kg | PRM-151 10 mg/kg | Total
Number analyzed (Participants) | 6 | 6 | 5 | 4 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.5 (12.88) | 63.7 (8.45) | 70.6 (8.26) | 66.5 (5.69) | 66.4 (9.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 1 | 0 | 4
  Male | 4 | 5 | 4 | 4 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 1
  White | 5 | 6 | 5 | 4 | 20
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 1 | 2 | 4 | 9
  Netherlands | 4 | 5 | 3 | 0 | 12
FVC [Mean (Standard Deviation); unit: liters] — Forced Vital Capacity: volume of air that can forcibly be blown out after full inspiration, measured in liters
  liters | 2.15 (0.64) | 2.96 (0.85) | 2.78 (0.73) | 2.97 (0.71) | 2.67 (0.76)
FVC % Predicted [Mean (Standard Deviation); unit: percent] — The % of the FVC that would be predicted for a subject based on physical characteristics that influence the maximal inhalation: height, age, and gender.
  percent | 63.2 (16.7) | 82.4 (15.5) | 80.0 (7.8) | 72.8 (14.3) | 74.1 (15.3)
FEV1 % Predicted [Mean (Standard Deviation); unit: percent] — Forced Expiratory Volume 1 second: the volume of air expired in the first second during maximal expiratory effort. FEV1% predicted is the FEV1% of the patient divided by the average FEV1% in the population for any person of similar age, sex and body composition
  percent | 68.8 (17.7) | 85.8 (16.8) | 87.0 (11.9) | 73.0 (12.1) | 78.5 (16.2)
DLCO [Mean (Standard Deviation); unit: percent] — Diffusing capacity carbon monoxide is the carbon monoxide uptake from a single inspiration in a standard time (usually 10 seconds). DLCO% predicted is the % of the DLCO that would be predicted based on the subject's hemoglobin.
  percent | 35.2 (8.4) | 41.2 (10.5) | 52.8 (9.8) | 46.0 (7.2) | 43.3 (10.9)

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability
Description: Number of subjects with Dose Limiting Toxicities, Number of Treatment Emergent Serious Adverse Events and Adverse Events
Time Frame: From first dose on Day 1 through Day 57
Population: All subjects who received at least one dose of study treatment
Measure: Number; unit: participants
Arm/Group | Placebo | PRM-151 1 mg/kg | PRM-151 5 mg/kg | PRM-151 10 mg/kg
Number analyzed (Participants) | 6 | 6 | 5 | 4
participants
  Dose Limiting Toxicities | 0 | 0 | 0 | 0
  Serious Adverse Events | 0 | 0 | 0 | 0
  Adverse Events | 6 | 6 | 5 | 4

2. Secondary Outcome: Cmax
Description: Maximum concentration
Time Frame: Day 15
Population: Subjects who received all doses of study treatment
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | PRM-151 1 mg/kg | PRM-151 5 mg/kg | PRM-151 10 mg/kg
Number analyzed (Participants) | 5 | 5 | 4
µg/mL | 25.5 (7.9) | 145 (41.9) | 225 (43.7)

3. Secondary Outcome: Tmax
Description: Time of Maximum observed concentration
Time Frame: Day 15
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | PRM-151 1 mg/kg | PRM-151 5 mg/kg | PRM-151 10 mg/kg
Number analyzed (Participants) | 5 | 5 | 4
hours | 5.35 (10.4) | 1.30 (1.51) | 0.69 (1.25)

4. Secondary Outcome: AUC48
Description: Area under the curve from 0 to 48 hrs post dose, with samples collected at 0.5, 0.75, 1, 1.5, 2, 3,4,6,8,12,16, 24 and 48 hours post Day 15 dose.
Time Frame: Day 15
Measure: Mean (Standard Deviation); unit: µg*hr/mL
Arm/Group | PRM-151 1 mg/kg | PRM-151 5 mg/kg | PRM-151 10 mg/kg
Number analyzed (Participants) | 5 | 5 | 4
µg*hr/mL | 446 (118) | 2190 (1140) | 4710 (1180)

5. Secondary Outcome: Terminal Elimination Half Life
Time Frame: Day 15
Measure: Mean (Full Range); unit: hour
Arm/Group | PRM-151 1 mg/kg | PRM-151 5 mg/kg | PRM-151 10 mg/kg
Number analyzed (Participants) | 5 | 5 | 4
hour | 21.7 [14.0 to 29.3] | 43.6 [11.2 to 79.2] | 71.6 [32.8 to 110.0]

6. Secondary Outcome: Total Body Clearance
Time Frame: Day 15
Measure: Mean (Full Range); unit: ml/hr/kg
Arm/Group | PRM-151 1 mg/kg | PRM-151 5 mg/kg | PRM-151 10 mg/kg
Number analyzed (Participants) | 5 | 5 | 4
ml/hr/kg | 2.33 [1.17 to 3.48] | 1.59 [0.780 to 2.65] | 1.09 [0.749 to 1.42]

7. Secondary Outcome: Vss
Description: Volume of Distribution at Steady State
Time Frame: Day 15
Measure: Mean (Full Range); unit: mL/kg
Arm/Group | PRM-151 1 mg/kg | PRM-151 5 mg/kg | PRM-151 10 mg/kg
Number analyzed (Participants) | 5 | 5 | 4
mL/kg | 53.9 [49.8 to 57.9] | 73.9 [37.6 to 139.0] | 72.0 [58.8 to 85.2]

8. Secondary Outcome: FVC (Forced Vital Capacity) Change From Baseline to Day 57
Time Frame: Change from Day 1 (Baseline) to Day 57
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Placebo | PRM-151 1 mg/kg | PRM-151 5 mg/kg | PRM-151 10 mg/kg
Number analyzed (Participants) | 6 | 5 | 5 | 4
liters | -0.063 (0.116) | 0.058 (0.164) | 0.060 (0.074) | 0.078 (0.210)

9. Secondary Outcome: FVC (Forced Vital Capacity) % Predicted Change From Baseline
Time Frame: Day 1 (Baseline) and Day 57
Measure: Mean (Standard Deviation); unit: absolute change in % predicted FVC
Arm/Group | Placebo | PRM-151 1 mg/kg | PRM-151 5 mg/kg | PRM-151 10 mg/kg
Number analyzed (Participants) | 6 | 5 | 5 | 4
absolute change in % predicted FVC | -1.5 (3.3) | 2.4 (4.6) | 2.8 (3.0) | 1.8 (5.3)

10. Secondary Outcome: DLCO (%) (Diffusing Capacity of Carbon Monoxide) Change From Baseline
Time Frame: Day 1 (Baseline) and Day 57
Measure: Mean (Standard Deviation); unit: Absolute change in % predicted DLCO
Arm/Group | Placebo | PRM-151 1 mg/kg | PRM-151 5 mg/kg | PRM-151 10 mg/kg
Number analyzed (Participants) | 6 | 5 | 5 | 4
Absolute change in % predicted DLCO | -2.3 (2.1) | 0.2 (3.3) | -4.0 (6.8) | -1.5 (3.8)

11. Secondary Outcome: FEV1 (Forced Expiratory Volume 1sec )(%) Change From Baseline
Time Frame: Day 1 (Baseline) and Day 57
Measure: Mean (Standard Deviation); unit: Absolute change in FEV1 % predicted
Arm/Group | Placebo | PRM-151 1 mg/kg | PRM-151 5 mg/kg | PRM-151 10 mg/kg
Number analyzed (Participants) | 6 | 5 | 5 | 4
Absolute change in FEV1 % predicted | -1.7 (4.3) | 2.6 (4.3) | 2.4 (1.1) | 0.3 (3.8)

12. Secondary Outcome: 6MWT (6 Minute Walk Test) Distance Walked Change From Baseline
Description: Change from baseline (measured during screening period) in distance walked during a 6 minute walk test
Time Frame: Screening (between Day -35 and Day 1) and Day 57
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Placebo | PRM-151 1 mg/kg | PRM-151 5 mg/kg | PRM-151 10 mg/kg
Number analyzed (Participants) | 6 | 5 | 5 | 4
meters | -11 (51) | -11 (63) | 6 (43) | 35 (45)

13. Secondary Outcome: SGRQ (St. George's Respiratory Questionnaire) Total Score Change From Baseline
Description: St. George's Respiratory Questionnaire Total Score. Scores range from 0 (no impairment) to 100 (maximum impairment). A decrease in score represents a decrease in disease related symptoms. The SGRQ is not validated for IPF.
Time Frame: Day 1 (Baseline) and Day 57
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | PRM-151 1 mg/kg | PRM-151 5 mg/kg | PRM-151 10 mg/kg
Number analyzed (Participants) | 6 | 5 | 5 | 4
units on a scale | -0.5 (6.2) | 2.3 (17.9) | 7.1 (12.0) | -6.3 (6.6)

ADVERSE EVENTS:
Arm/Group | Placebo | PRM-151 1 mg/kg | PRM-151 5 mg/kg | PRM-151 10 mg/kg
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/5 | 0/4
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 5/5 | 4/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=6) | PRM-151 1 mg/kg (N=6) | PRM-151 5 mg/kg (N=5) | PRM-151 10 mg/kg (N=4)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 3 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2 | 1
Fatigue (General disorders) | 1 | 0 | 2 | 1
Headache (Nervous system disorders) | 1 | 2 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0
Hematoma (General disorders) | 1 | 2 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 2 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0
Catheter site hematoma (General disorders) | 1 | 1 | 0 | 0
Malaise (General disorders) | 1 | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 2 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators agree that the first public presentation of data will be a joint, multicentre publication of results. If this does not occur within 12 months after conclusion of the study, investigator may publish the results, provided that the complete manuscript or other publication is submitted to the sponsor for review 30 days prior to submission.